CLINICAL TRIAL: NCT03924453
Title: Use and Effectiveness of a Digitally Integrated Ovulation Prediction Kits for Fertility Tracking - Pearl Powered by Proov
Brief Title: Usability Study of the Pearl Fertility Tracking Device
Status: Completed | Type: Observational
Sponsor: MFB Fertility (Industry)
Responsible Party: Sponsor
Other Study IDs: 2017/11/7
Record Dates: First submitted 2019-04-17; First posted 2019-04-23 (Actual); Last update posted 2020-09-03 (Actual); Status verified 2020-09

CONDITIONS: Ovulation Disorder

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pearl Powered by Proov: Participants are given hormone tests strips and a digital app and all instructions for use, collectively called the Pearl Power by Proov kit. The app will analyze hormonal test strip information to predict and confirm ovulation
  Interventions: Diagnostic Test: Pearl Powered by Proov

INTERVENTIONS:
Diagnostic Test: Pearl Powered by Proov — Participants self test in their homes and report back data via uploading onto an app and taking surveys.

SUMMARY:
This mobile application measures the level of certain hormones in the urine of a woman and is used to help pinpoint when the woman is/was most likely to get pregnant during her menstrual cycle.

DETAILED DESCRIPTION:
The purpose of the study is to evaluate the accuracy of ovulation monitoring using hormone test strips in a digital way via a mobile application.

Ovulation prediction kits consist of test strips that measure three different hormones - LH (luteinizing hormone), FSH (follicle stimulating hormone), PdG (pregnanediol). Through daily testing with the mobile application, it is possible to measure these hormones and build hormonal profiles along the menstrual cycle. This way we can accurately predict and confirm ovulation, as well as calculate the most fertile days in the cycle.

There are multiple solutions that claim to accurately monitor fertility. However, some of these solutions use period statistics with high level of error, for example period trackers, or body temperature monitors. Some others use hormonal test strips in which reading/interpretation is not always easy. This study evaluates the accuracy of using hormone test strips in combination with an app that will digitally read and record data over time.

ELIGIBILITY:
Inclusion Criteria:

1. Female (mandatory)
2. Not currently pregnant or nursing (mandatory)
3. Aged 21-45 (advanced age can hinder hormone levels)
4. Not be diagnosed as sub fertile (infertility causes inconsistent hormone levels)
5. Not have used any form of hormonal birth control in the past 2 months (mandatory)
6. Currently trying to conceive (ideal but not required)
7. Currently reside in the US (mandatory, this study is for US residents only)

Exclusion Criteria:

1. Male
2. Pregnant
3. Nursing

Ages: 18 Years to 45 Years | Sex: Female
Age Groups: Adult
Gender Based: Yes — female only due to ovulation tracking diagnostic
Study Population: Women aged 18-45 that are activity seeking to get pregnant and want to monitor their fertility status
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Number of Participants with positive PDG test results | A single menstrual cycle, up to 45 days
  phone application will be used to record LH, FSH, and PDG tests. Number of participants with positive PDG test strips will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Amy Beckley, PhD, Principal Investigator — MFB Fertility
Locations (1):
- MFB Fertility, Boulder, Colorado, United States

IPD SHARING:
Plan to Share IPD: No